CLINICAL TRIAL: NCT01023958
Title: An Open-label, Single-arm, Phase II Trial of Intravenous BI 6727 in Patients With Locally Advanced, Metastatic or Recurrent Urothelial Cancer of the Bladder, Renal Pelvis, or Ureters After Failure of Prior Chemotherapy
Brief Title: Intravenous BI 6727 (Volasertib) in 2nd Line Treatment of Urothelial Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1230.2
Record Dates: First submitted 2009-11-24; First posted 2009-12-02 (Estimated); Results first posted 2017-11-22 (Actual); Last update posted 2017-11-22 (Actual); Status verified 2017-10

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — BI 6727; Infusions, Intravenous

ARMS (1):
- single arm (Experimental): open label
  Interventions: Drug: BI 6727, IV infusion

INTERVENTIONS:
Drug: BI 6727, IV infusion — phase II

SUMMARY:
The primary objective of this trial is to evaluate the efficacy and safety of BI 6727 in patients with locally advanced, metastatic or recurrent urothelial cancer after failure of first line or adjuvant/neoadjuvant chemotherapy.

ELIGIBILITY:
Inclusion criteria:

1. Histologically or cytologically confirmed urothelial cancer of the bladder, ureters or renal pelvis.
2. Patients with stage III, IV or recurrent urothelial cancer of the bladder, ureter or renal pelvis after failure or recurrence after first line or adjuvant/neoadjuvant chemotherapy. Recurrence is defined as relapse within 2 years after cessation of prior first-line chemotherapy.
3. Male or female patient aged 18 years or older
4. Life expectancy of at least three (3) months
5. Eastern Co-operative Oncology Group performance score of 2 or less
6. At least one target tumor lesion that has not been irradiated within the past three months and that can accurately be measured by magnetic resonance imaging (MRI) or computed tomography (CT) in at least one dimension (longest diameter to be recorded) as >20 mm with conventional techniques or as >10 mm with spiral CT
7. The patient must have given written informed consent prior to inclusion into the trial which must be consistent with the International Conference on Harmonization, Good Clinical Practice (ICH-GCP) and local legislation

Exclusion criteria:

1. More than one prior regimen of chemotherapy including prior adjuvant therapy
2. Brain metastases
3. Patients with bone metastasis as the only site of disease are excluded
4. Serious illness or organ system dysfunction, which in the opinion of the investigator, would either compromise patient safety, interfere with the evaluation of the safety of the test drug or limit compliance with trial requirements.
5. QTc prolongation deemed clinically relevant by the investigator
6. Second malignancy currently requiring active therapy
7. Other active malignancy diagnosed within the past 3 years (other than non melanomatous skin cancer and cervical intraepithelial neoplasia)
8. Absolute neutrophil count (ANC) <1,500/µl
9. Platelet count <100,000/µl
10. Hemoglobin <9 g/dl
11. Total bilirubin >1.5 mg/dl
12. Aspartate amino transferase (AST) and/or alanine amino transferase (ALT) >2.5 x ULN, or aspartate amino transferase (AST) and/or alanine amino transferase (ALT) >5 x ULN in case of known liver metastases
13. Serum creatinine >1.5 x ULN
14. Chemo-, Radio- or immunotherapy within the past 4 weeks. This does not apply to steroids and bisphosphonates.
15. Active infectious disease, or HIV, Hepatitis-B or -C infection
16. Active drug or alcohol abuse
17. Women and men who are sexually active and unwilling to use a medically acceptable method of contraception (e.g. such as implants, injectables, combined oral contraceptives, some intrauterine devices or vasectomized partner for participating females, condoms for participating males) during the trial
18. Pregnancy or breast feeding
19. Treatment with any investigational drug within the past 4 weeks or within less than four half-life times of the investigational drug before treatment with the trial drug and/or persistence of toxicities of prior anticancer therapies which are deemed to be clinically relevant.
20. Prior treatment with Polo-like kinase 1 (Plk1) inhibitor
21. Patient unable to comply with the protocol
22. Any known hypersensitivity to the trial drugs or their excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-11-19 (Actual); Primary Completion 2011-09-19 (Actual); Study Completion 2011-09-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (21):
- United States (19):
  - 1230.2.5 Boehringer Ingelheim Investigational Site, Beverly Hills, California
  - 1230.2.10 Boehringer Ingelheim Investigational Site, Los Angeles, California
  - 1230.2.34 Boehringer Ingelheim Investigational Site, Miami, Florida
  - 1230.2.29 Boehringer Ingelheim Investigational Site, Orlando, Florida
  - 1230.2.6 Boehringer Ingelheim Investigational Site, Chicago, Illinois
  - 1230.2.17 Boehringer Ingelheim Investigational Site, Joliet, Illinois
  - 1230.2.24 Boehringer Ingelheim Investigational Site, Metairie, Louisiana
  - 1230.2.1 Boehringer Ingelheim Investigational Site, Baltimore, Maryland
  - 1230.2.25 Boehringer Ingelheim Investigational Site, Las Vegas, Nevada
  - 1230.2.36 Boehringer Ingelheim Investigational Site, Las Vegas, Nevada
  - 1230.2.19 Boehringer Ingelheim Investigational Site, Lebanon, New Hampshire
  - 1230.2.20 Boehringer Ingelheim Investigational Site, New York, New York
  - 1230.2.23 Boehringer Ingelheim Investigational Site, New York, New York
  - 1230.2.12 Boehringer Ingelheim Investigational Site, Charlotte, North Carolina
  - 1230.2.4 Boehringer Ingelheim Investigational Site, Philadelphia, Pennsylvania
  - 1230.2.38 Boehringer Ingelheim Investigational Site, Beaumont, Texas
  - 1230.2.41 Boehringer Ingelheim Investigational Site, Tyler, Texas
  - 1230.2.43 Boehringer Ingelheim Investigational Site, Webster, Texas
  - 1230.2.44 Boehringer Ingelheim Investigational Site, Fairfax, Virginia
- Taiwan (2):
  - 1230.2.51 Boehringer Ingelheim Investigational Site, Tainan
  - 1230.2.50 Boehringer Ingelheim Investigational Site, Taipei

REFERENCES:
- [Derived] Stadler WM, Vaughn DJ, Sonpavde G, Vogelzang NJ, Tagawa ST, Petrylak DP, Rosen P, Lin CC, Mahoney J, Modi S, Lee P, Ernstoff MS, Su WC, Spira A, Pilz K, Vinisko R, Schloss C, Fritsch H, Zhao C, Carducci MA. An open-label, single-arm, phase 2 trial of the Polo-like kinase inhibitor volasertib (BI 6727) in patients with locally advanced or metastatic urothelial cancer. Cancer. 2014 Apr 1;120(7):976-82. doi: 10.1002/cncr.28519. Epub 2013 Dec 11. PMID 24339028

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: An open-label, single-arm, Phase II trial of intravenous volasertib (BI 6727) in patients with locally advanced, metastatic or recurrent urothelial cancer of the bladder, renal pelvis, or ureters after failure of prior chemotherapy.
Groups:
- Volasertib (BI 6727): Volasertib (BI 6727) was administered as intravenous infusion over 2 hours at Day 1 of each 21-day treatment course. Single dose, 300 mg as starting dose in first treatment course - possible dose escalation at the beginning of the 2nd course to 350 mg if well tolerated. Repeated administration in patients with clinical benefit until disease progression or intolerability of the study medication
Period: Overall Study
Arm/Group | Volasertib (BI 6727)
Started | 50
Completed | 0
Not Completed | 50
Not completed — Progressive disease | 48
Not completed — Other adverse event | 1
Not completed — Refused to continue medication | 1

BASELINE CHARACTERISTICS:
Population: Treated set (TS) which included all patients who received at least one dose of trial medication.
Arm/Group | Volasertib (BI 6727)
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: Years] | 69.0 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 40

OUTCOME MEASURES:

1. Primary Outcome: Objective Tumour Response According to RECIST Criteria
Description: Objective tumor response, defined as complete response (CR) or partial response (PR), according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria.
Time Frame: From first drug administration until end of study, up to 2 years
Population: TS
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Volasertib (BI 6727)
Number analyzed (Participants) | 50
Percentage of participants | 14.0 [5.8 to 26.7]

2. Secondary Outcome: Progression-free Survival
Description: Progression-free survival (PFS) is the time from first treatment to the occurrence of tumor progression or death, whichever occurs first. Disease progression is defined according to the RECIST guideline but also includes the investigators' assessment which may, in some cases, include only clinical progression (deterioration of general health status per investigator). PFS was analyzed with the Kaplan-Meier curve. Greenwood's variance estimate was used to form confidence intervals.
  Patients without evidence of disease progression were to be censored at the last image date.
Time Frame: Time from first treatment to the occurrence of tumor progression or death, up to 2 years
Population: TS
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Volasertib (BI 6727)
Number analyzed (Participants) | 50
Weeks | 6.1 [5.6 to 11.1]

3. Secondary Outcome: Overall Survival
Description: Overall survival (OS) is the time from first infusion to death. Patients who were alive at the time of analysis or lost to follow-up were censored at the last follow-up date when they were known to be alive.
  Overall survival was analyzed with the Kaplan-Meier curve. Greenwood's variance estimate was used to form confidence intervals.
Time Frame: Time from first infusion to death, up to 2 years
Population: TS
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Volasertib (BI 6727)
Number analyzed (Participants) | 50
Months | 8.5 [3.9 to 12.1]

4. Secondary Outcome: Duration of Overall Response
Description: The duration of overall response is measured from the time of first response (CR or PR) to progression or death whichever occurs first.
Time Frame: From the time of first response (CR or PR) to progression or death, up to 2 years
Population: TS
Measure: Median (Full Range); unit: Weeks
Arm/Group | Volasertib (BI 6727)
Number analyzed (Participants) | 7
Weeks | 41.0 [29.1 to 77.3]

5. Secondary Outcome: Disease Control Rate
Description: Disease control rate. Disease control is defined as having a best overall response of complete response (CR), partial response (PR) or stable disease (SD).
Time Frame: From first drug administration until end of study, up to 2 years
Population: TS
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Volasertib (BI 6727)
Number analyzed (Participants) | 50
Percentage of participants | 40.0 [26.4 to 54.8]

6. Secondary Outcome: Duration of Disease Control
Description: Disease control is defined as having a best overall response of CR, PR, or SD. The duration of disease control is measured from the time of first response to progression or death whichever occurs first.
Time Frame: Time of first response to progression or death, up to 2 years
Population: Patients who achieved disease control in the TS.
Measure: Median (Full Range); unit: Weeks
Arm/Group | Volasertib (BI 6727)
Number analyzed (Participants) | 20
Weeks | 27.0 [10.1 to 77.3]

7. Secondary Outcome: AUC0-∞ of Volasertib
Description: Area under the concentration-time curve in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) of volasertib
Time Frame: 5 mins before start of drug infusion and 2h, 3h, 6h, 24h, 168h and 336h after start of drug infusion
Population: Pharmacokinetic set (PKS) including patients with analyzable data for this endpoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Volasertib (BI 6727)
Number analyzed (Participants) | 48
ng*h/mL | 5470 (30.6)

8. Secondary Outcome: Cmax of Volasertib
Description: Maximum measured concentration in plasma (Cmax) of volasertib
Time Frame: 5 mins before start of drug infusion and 2h, 3h, 6h, 24h, 168h and 336h after start of drug infusion
Population: PKS including patients with analyzable data for this endpoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Volasertib (BI 6727)
Number analyzed (Participants) | 47
ng/mL | 253 (51.9)

9. Secondary Outcome: t1/2 of Volasertib
Description: Terminal half-life (t1/2) of volasertib
Time Frame: 5 mins before start of drug infusion and 2h, 3h, 6h, 24h, 168h and 336h after start of drug infusion
Population: PKS including patients with analyzable data for this endpoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Volasertib (BI 6727)
Number analyzed (Participants) | 48
hours | 150 (17.0)

10. Secondary Outcome: CL of Volasertib
Description: Total plasma clearance after intravascular administration (CL) of volasertib
Time Frame: 5 mins before start of drug infusion and 2h, 3h, 6h, 24h, 168h and 336h after start of drug infusion
Population: PKS including patients with analyzable data for this endpoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min
Arm/Group | Volasertib (BI 6727)
Number analyzed (Participants) | 48
mL/min | 914 (30.6)

11. Secondary Outcome: Vss of Volasertib
Description: Apparent volume of distribution at steady state following intravascular administration (Vss) of volasertib
Time Frame: 5 mins before start of drug infusion and 2h, 3h, 6h, 24h, 168h and 336h after start of drug infusion
Population: PKS including patients with analyzable data for this endpoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Litres
Arm/Group | Volasertib (BI 6727)
Number analyzed (Participants) | 48
Litres | 7470 (32.4)

12. Secondary Outcome: Tmax of Volasertib
Description: Time from dosing to maximum measured concentration (Tmax) of volasertib
Time Frame: 5 mins before start of drug infusion and 2h, 3h, 6h, 24h, 168h and 336h after start of drug infusion
Population: PKS including patients with analyzable data for this endpoint.
Measure: Median (Full Range); unit: Hours
Arm/Group | Volasertib (BI 6727)
Number analyzed (Participants) | 47
Hours | 2.03 [1.53 to 4.17]

13. Secondary Outcome: Occurrence and Intensity of AE's Graded According to CTCAE
Description: Occurrence and intensity of adverse events (AEs) graded according to Common Toxicity Criteria of Adverse Events (CTCAE).
  The CTCAE grades are: 1 (mild AE), 2 (moderate AE), 3 (severe AE), 4 (life-threatening or disabling AE), 5 (death related to AE).
Time Frame: From first drug administration until end of study, up to 2 years
Population: TS
Measure: Number; unit: Percentage of participants
Arm/Group | Volasertib (BI 6727)
Number analyzed (Participants) | 50
Percentage of participants
  Grade 1 | 8.0
  Grade 2 | 28.0
  Grade 3 | 36.0
  Grade 4 | 20.0
  Grade 5 | 6.0

14. Secondary Outcome: Occurrence of Unacceptable Toxicity
Description: Occurrence of unacceptable toxicity is defined by CTCAE as as drug related CTCAE Grade 3 or greater non-hematological toxicity (except emesis or diarrhea responding to supportive treatment); drug-related CTCAE Grade 4 neutropenia for seven or more days and / or complicated by infection; or drug-related CTCAE Grade 4 thrombocytopenia.
Time Frame: From first drug administration up to 21 days after final administration, up to 2 years
Population: TS
Measure: Number; unit: Percentage of participants
Arm/Group | Volasertib (BI 6727)
Number analyzed (Participants) | 50
Percentage of participants | 30

15. Secondary Outcome: Laboratory Investigation: Haemoglobin
Description: Difference from baseline in laboratory parameter Haemoglobin
Time Frame: Baseline and last value on treatment (up to 2 years)
Population: TS. Results displayed for patients with available haemoglobin data.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Volasertib (BI 6727)
Number analyzed (Participants) | 49
g/L | -19 (24)

16. Secondary Outcome: Laboratory Investigation: White Blood Cell Count
Description: Difference from baseline in laboratory parameter white blood cell count
Time Frame: Baseline and last value on treatment (up to 2 years)
Population: TS. Results displayed for patients with available white blood cell count data.
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Volasertib (BI 6727)
Number analyzed (Participants) | 49
10^9 cells/L | -1.8 (4.0)

17. Secondary Outcome: Laboratory Investigation: Platelets
Description: Difference from baseline in laboratory parameter Platelets
Time Frame: Baseline and last value on treatment (up to 2 years)
Population: TS. Results displayed for patients with available platelets data.
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Volasertib (BI 6727)
Number analyzed (Participants) | 49
10^9 cells/L | -23 (89)

18. Secondary Outcome: Laboratory Investigation: Neutrophils
Description: Difference from baseline in laboratory parameter Neutrophils
Time Frame: Baseline and last value on treatment (up to 2 years)
Population: TS. Results displayed for patients with available neutrophils data.
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Volasertib (BI 6727)
Number analyzed (Participants) | 49
10^9 cells/L | -1.9 (6.3)

19. Secondary Outcome: Laboratory Investigation: Lymphocytes
Description: Difference from baseline in laboratory parameter Lymphocytes
Time Frame: Baseline and last value on treatment (up to 2 years)
Population: TS. Results displayed for patients with available lymphocytes data.
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Volasertib (BI 6727)
Number analyzed (Participants) | 49
10^9 cells/L | -0.8 (4.0)

20. Secondary Outcome: Laboratory Investigation: AST/GOT, SGOT
Description: Difference from baseline in laboratory parameter Aspartate aminotransferase(AST)/GOT, SGOT
Time Frame: Baseline and last value on treatment (up to 2 years)
Population: TS. Results displayed for patients with available AST/GOT, SGOT data.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Volasertib (BI 6727)
Number analyzed (Participants) | 49
U/L | 5 (26)

21. Secondary Outcome: Laboratory Investigation: ALT/GPT, SGPT
Description: Difference from baseline in laboratory parameter Alanine aminotransferase(ALT)/GPT, SGPT
Time Frame: Baseline and last value on treatment (up to 2 years)
Population: TS. Results displayed for patients with available ALT/GPT, SGPT data.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Volasertib (BI 6727)
Number analyzed (Participants) | 49
U/L | 3 (19)

22. Secondary Outcome: Laboratory Investigation: Alkaline Phosphatase
Description: Difference from baseline in laboratory parameter Alkaline phosphatase
Time Frame: Baseline and last value on treatment (up to 2 years)
Population: TS. Results displayed for patients with available alkaline phosphate data.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Volasertib (BI 6727)
Number analyzed (Participants) | 49
U/L | 35 (95)

23. Secondary Outcome: Laboratory Investigation: Creatinine
Description: Difference from baseline in laboratory parameter Creatinine
Time Frame: Baseline and last value on treatment (up to 2 years)
Population: TS. Results displayed for patients with available creatinine data.
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Volasertib (BI 6727)
Number analyzed (Participants) | 49
umol/L | 16 (41)

24. Secondary Outcome: Laboratory Investigation: Total Bilirubin
Description: Difference from baseline in laboratory parameter total Bilirubin
Time Frame: Baseline and last value on treatment (up to 2 years)
Population: TS. Results displayed for patients with available total bilirubin data.
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Volasertib (BI 6727)
Number analyzed (Participants) | 49
umol/L | 4.7 (34.1)

ADVERSE EVENTS:
Time Frame: From first drug administration until end of study, up to 2 years
Arm/Group | Volasertib (BI 6727)
Serious Adverse Events (participants affected / at risk) | 13/50
Other Adverse Events (participants affected / at risk) | 49/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Volasertib (BI 6727) (N=50)
Anaemia (Blood and lymphatic system disorders) | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 1
Pyrexia (General disorders) | 1
Bacteraemia (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Perirectal abscess (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 2
Urosepsis (Infections and infestations) | 1
Foreign body (Injury, poisoning and procedural complications) | 1
Urostomy complication (Injury, poisoning and procedural complications) | 1
Decreased appetite (Metabolism and nutrition disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 2
Hyponatraemia (Metabolism and nutrition disorders) | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Convulsion (Nervous system disorders) | 1
Confusional state (Psychiatric disorders) | 1
Mental status changes (Psychiatric disorders) | 1
Renal failure acute (Renal and urinary disorders) | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Volasertib (BI 6727) (N=50)
Anaemia (Blood and lymphatic system disorders) | 20
Leukopenia (Blood and lymphatic system disorders) | 5
Neutropenia (Blood and lymphatic system disorders) | 15
Thrombocytopenia (Blood and lymphatic system disorders) | 19
Abdominal pain (Gastrointestinal disorders) | 3
Abdominal pain lower (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 16
Diarrhoea (Gastrointestinal disorders) | 11
Nausea (Gastrointestinal disorders) | 19
Vomiting (Gastrointestinal disorders) | 6
Asthenia (General disorders) | 5
Chest pain (General disorders) | 3
Chills (General disorders) | 3
Fatigue (General disorders) | 28
Oedema peripheral (General disorders) | 4
Pain (General disorders) | 3
Pyrexia (General disorders) | 5
Oral candidiasis (Infections and infestations) | 3
Urinary tract infection (Infections and infestations) | 6
Blood creatinine increased (Investigations) | 3
Weight decreased (Investigations) | 4
Decreased appetite (Metabolism and nutrition disorders) | 16
Dehydration (Metabolism and nutrition disorders) | 6
Hypercalcaemia (Metabolism and nutrition disorders) | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 3
Hyponatraemia (Metabolism and nutrition disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 11
Groin pain (Musculoskeletal and connective tissue disorders) | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4
Dizziness (Nervous system disorders) | 7
Anxiety (Psychiatric disorders) | 6
Depression (Psychiatric disorders) | 4
Insomnia (Psychiatric disorders) | 6
Dysuria (Renal and urinary disorders) | 4
Pollakiuria (Renal and urinary disorders) | 4
Renal failure (Renal and urinary disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 10
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7
Alopecia (Skin and subcutaneous tissue disorders) | 4
Rash (Skin and subcutaneous tissue disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.